CLINICAL TRIAL: NCT04400396
Title: Effect of Target vs. Standard Human Milk Fortification on the Growth and Body Composition of Predominantly Human Milk Fed Very Preterm Infants
Brief Title: Effect of Target Fortified Human Milk on the Growth Quality of Very Preterm Infants (TargetFort)
Acronym: TargetFort
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Centro Hospitalar de Lisboa Central (Other)
Collaborators: Sociedade Portuguesa de Neonatologia (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHULC.CI512.2020
Record Dates: First submitted 2020-05-18; First posted 2020-05-22 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Growth; Body Composition; Prematurity; Breast Milk Collection; Nutrient Deficiency; Feeding Patterns; Adiposity
MeSH Terms: conditions — Premature Birth; Breast Milk Expression; Feeding Behavior; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Human milk (HM), including mother's own milk (MOM) and donor's milk (DHM).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- target HM fortification: Contemporary cohort fed HM with target fortification
  Interventions: Dietary Supplement: target HM fortification
- standard HM fortification: Historical cohort fed HM with standard fortification
  Interventions: Dietary Supplement: standard HM fortification

INTERVENTIONS:
Dietary Supplement: standard HM fortification — Based on the assumed energy and macronutrient composition of HM, the commercial multi-component HM fortifier was added, in order to compensate identified nutritional deficits.
  Groups: standard HM fortification
Dietary Supplement: target HM fortification — Based on the measured energy and macronutrient composition of HM, modular protein and fat supplements are added, in addition to the commercial multi-component HM fortifier, in order to correct identified specific nutritional deficits. For this purpose, an Excel program to calculate modular protein and fat supplements to be added to fortified HM was developed and registered (Nona R, Cardoso M, Portuguese Directorate of Intellectual Property Services, IGAC-DSPI, nº 480/2020, 26 February 2020)
  Groups: target HM fortification

SUMMARY:
It is reported that the standard method for fortification of human milk (HM) overestimates the energy and protein densities of HM (Macedo MHNP 2018), thus originating infant undernutrition (Macedo AJP 2018). The target fortification, based on analysis of HM composition, is considered the gold-standard method (Rochow 2015, McLeod 2016). This observational mixed cohort study aims to assess if very preterm infants fed HM with target fortification have greater growth during hospital stay and better body composition at term post-menstrual age (PMA), than those fed HM with standard fortification.

DETAILED DESCRIPTION:
Study design: observational mixed cohort study, comparing growth and body composition in a contemporary cohort of very preterm infants fed HM with target fortification, the currently adopted clinical practice, with a historical cohort of very preterm infants fed HM with standard fortification (Macedo AJP 2018).

Study periods: historical cohort from 1 February 2014 to 28 February 2015; contemporary cohort: start February 2020, estimated recruitment period of 16 months; Settings: Neonatal Care Unit (NICU) and Human Milk Bank at Maternidade Dr. Alfredo da Costa and Nutrition Laboratory at Hospital Dona Estefânia, Centro Hospitalar Universitário de Lisboa Central.

Product to be analyzed: HM, including mother's own milk (MOM) and donor's milk (DHM). Donor HM is pasteurized using the Holder method (Peila 2016) which is adopted by the Human Milk Bank of Maternidade Dr. Alfredo da Costa (Macedo MHNP 2018).

Demographic variables: Gestational age, sex, singleton or twin, birth weight, small-, appropriate- or large-for-gestational age (<3rd percentile, ≥3rd percentile and ≤97th percentile, >97th percentile, respectively) (Fenton 2013), severity index (SNAPPE II) (Richardson 2001), use of prenatal corticosteroids, diagnosis of late sepsis (Modi 2009), necrotizing enterocolitis (grade ≥ 3) (Bell 1971), intraperiventricular hemorrhage (grade ≥ 3) (Papile 1978), multicystic periventricular leukomalacia (de Vries 1992), and chronic lung disease (Becker 1984).

Method of collection and analysis of HM: as described in a previous study (Macedo MHNP 2018), in order to minimize daily variability of breast milk composition, mothers are asked to save milk collected through 24 hours in the same container. The HM composition (MOM and DHM) are analyzed using the Miris human milk analyzer (Miris AB, Uppsala, Sweden), following the method described in a previous study (Macedo MHNP 2018). The composition is expressed in densities: Kcal/dL of energy and g/dl of fat, raw and true protein, carbohydrates and ashes.

Energy and macronutrient composition of the multi-component HM fortifier and modular protein and fat supplements. For this purpose, an Excel program to calculate modular protein and fat supplements to be added to fortified HM was developed and registered (Nona R, Cardoso M, Portuguese Directorate of Intellectual Property Services, IGAC-DSPI, nº 480/2020, 26 February 2020).

Daily intakes of energy (Kcal/kg), protein (g/kg) and protein:energy ratio (P:E), based on administered volume of milk (ml/kg).

Anthropometric and body composition measurements in infants: According to the previously described method (Macedo AJP 2018), during the hospital stay, the same observer (MMC) measures daily the body weight (allowing the calculation of weight gain velocity), and weekly the length and the head circumference. Within the first week after discharge, body composition will be assessed using displacement plethysmography, to evaluate fat mass (FM), fat free mass (FFM), percentage of FM (%FM), percentage of FFM (%FFM) and FM index (FMI), as described in a previous study (Macedo AJP 2018). Both FMI and %FM are used as indicators of adiposity.

Estimate of sample size: The study sample size was calculated to detect a difference of 2 g/kg/day in growth velocity with a standard deviation 2.6 (Macedo, 2018; Tremblay, 2017) for normally distributed variables, a significance level of 0.05, and an 80% power; thus, a required sample of 67 infants (n1=33; n2+20%=34) was estimated.

ELIGIBILITY:
Inclusion Criteria:

* newborn infants born at <33 weeks of gestation,
* admitted to the NICU of Maternidade Dr. Alfredo da Costa (inborns and outborns),
* exclusively or predominantly HM fed (>87.5% volume per day)
* discharged alive.

Exclusion Criteria:

* multiples of grade >2
* diagnosis of innate metabolism disorder,
* fed with formula for >12.5% of the daily volume intake for two or more consecutive full days ,
* discharge with transference to other hospital,
* unavailable for body composition analysis after discharge.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Very preterm newborn infants (born at <33 weeks) that achieve full enteral feeding exclusively or predominantly with human milk
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-16 (Estimated)

PRIMARY OUTCOMES:
weight gain velocity rate | from baseline (the first day of exclusive or predominantly feeding with fortified human milk) up to 40 weeks postmenstrual age or to home discharge, whatever comes first
  average relative daily variation of body weight
length velocity rate | from baseline (the first day of exclusive or predominantly feeding with fortified human milk) up to 40 weeks postmenstrual age or to home discharge, whatever comes first
  average relative weekly variation of body length
head circumference velocity rate | from baseline (the first day of exclusive or predominantly feeding with fortified human milk) up to 40 weeks postmenstrual age or to home discharge, whatever comes first
  average relative weekly variation of head circumference
adiposity (fat mass index) | A single measurement performed up to 10 days after home discharge
  ratio of fat mass over squared body length

SECONDARY OUTCOMES:
adiposity (fat mass percentage) | A single measurement performed up to 10 days after home discharge
  proportion of fat mass on total body mass

CONTACTS AND LOCATIONS:
Overall Officials: Luis Pereira-da-Silva, MD, PhD, Study Director — Universidade Nova de Lisboa
Locations (1):
- Centro Hospitalar Universitário de Lisboa Central, Lisbon, Portugal

REFERENCES:
- [Background] Macedo I, Pereira-da-Silva L, Cardoso M. The fortification method relying on assumed human milk composition overestimates the actual energy and macronutrient intakes in very preterm infants. Matern Health Neonatol Perinatol. 2018 Sep 17;4:22. doi: 10.1186/s40748-018-0090-4. eCollection 2018. PMID 30237896
- [Background] McLeod G, Sherriff J, Hartmann PE, Nathan E, Geddes D, Simmer K. Comparing different methods of human breast milk fortification using measured v. assumed macronutrient composition to target reference growth: a randomised controlled trial. Br J Nutr. 2016 Feb 14;115(3):431-9. doi: 10.1017/S0007114515004614. Epub 2015 Dec 2. PMID 26627899
- [Background] Rochow N, Landau-Crangle E, Fusch C. Challenges in breast milk fortification for preterm infants. Curr Opin Clin Nutr Metab Care. 2015 May;18(3):276-84. doi: 10.1097/MCO.0000000000000167. PMID 25807355
- [Result] Macedo I, Pereira-da-Silva L, Cardoso M. Associations of Measured Protein and Energy Intakes with Growth and Adiposity in Human Milk-Fed Preterm Infants at Term Postmenstrual Age: A Cohort Study. Am J Perinatol. 2018 Jul;35(9):882-891. doi: 10.1055/s-0038-1626717. Epub 2018 Feb 2. PMID 29532450
- [Result] Henriksen C, Westerberg AC, Ronnestad A, Nakstad B, Veierod MB, Drevon CA, Iversen PO. Growth and nutrient intake among very-low-birth-weight infants fed fortified human milk during hospitalisation. Br J Nutr. 2009 Oct;102(8):1179-86. doi: 10.1017/S0007114509371755. Epub 2009 May 18. PMID 19445820
- [Result] Maas C, Wiechers C, Bernhard W, Poets CF, Franz AR. Early feeding of fortified breast milk and in-hospital-growth in very premature infants: a retrospective cohort analysis. BMC Pediatr. 2013 Nov 4;13:178. doi: 10.1186/1471-2431-13-178. PMID 24180239
- [Result] Morlacchi L, Mallardi D, Gianni ML, Roggero P, Amato O, Piemontese P, Consonni D, Mosca F. Is targeted fortification of human breast milk an optimal nutrition strategy for preterm infants? An interventional study. J Transl Med. 2016 Jul 1;14(1):195. doi: 10.1186/s12967-016-0957-y. PMID 27370649
- [Result] Polberger S. New approaches to optimizing early diets. Nestle Nutr Workshop Ser Pediatr Program. 2009;63:195-204; discussion 204-8, 259-68. doi: 10.1159/000209982. PMID 19346777
- [Derived] Cardoso M, Virella D, Macedo I, Silva D, Pereira-da-Silva L. Customized Human Milk Fortification Based on Measured Human Milk Composition to Improve the Quality of Growth in Very Preterm Infants: A Mixed-Cohort Study Protocol. Int J Environ Res Public Health. 2021 Jan 19;18(2):823. doi: 10.3390/ijerph18020823. PMID 33477964